CLINICAL TRIAL: NCT05209971
Title: Macular Thickness and Visual Acuity in Diabetic Hypertensive Patients in Sohag City
Brief Title: Macular Thickness and Visual Acuity in Diabetic Hypertensive Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Raghda Abdelraheem Abdellah, principal investigator, Sohag University
Other Study IDs: Soh-Med-22-01-05
Record Dates: First submitted 2022-01-13; First posted 2022-01-27 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Macular Edema
Keywords: Macular thickness and visual acuity
MeSH Terms: conditions — Macular Edema

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- macular thickness and visual acuity: optical coherence tomography

SUMMARY:
In this study, measurements of central macular thickness using optical coherence tomography along with examination of visual acuity by Snellen's chart in diabetic hypertensive patients will be done .

DETAILED DESCRIPTION:
correlate relationship between optical coherence tomography changes and visual acuity in patients with type 2 diabetes and hypertension

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic patients with hypertension .

Exclusion Criteria:

* Patients with type 1 diabetes mellitus .
* Ocular disease ( such as high myopia , glaucoma ) .
* Patients with opacities in the media ( corneal opacities , dense cataract , vitreous hemorrhage ) .
* Systemic medication (Tamoxifen , Chloroquine , Canthaxanthine ) to avoid its effect on macular thickness .
* Central visual field defect that prevents fixation on OCT .
* Intraocular inflammation such as anterior or posterior uveitis .
* Refractive error greater than 6 diopter .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a retrospective study of patients of type 2 diabetes with hypertension
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
macular thickness in diabetic hypertensive patients | June 2022
  measurement of central macular thickness by optical coherence tomography

CONTACTS AND LOCATIONS:
Overall Officials: Raghda Abdelraheem, doctor, Principal Investigator — faculty of medicine

IPD SHARING:
Plan to Share IPD: No
measurement of macular thickness